CLINICAL TRIAL: NCT01532297
Title: Application of Citrate Dialysate in Chronic Haemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HD-CiDi-01-D; There is no secondary ID
Record Dates: First submitted 2011-10-20; First posted 2012-02-14 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Renal Disease
Keywords: citrate dialysate; dialysis; calcium
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- HD treated with standard dialysate (Active Comparator)
  Interventions: Device: Standard dialysate (StDi)
- post-dilution oHDF with standard dialysate (Active Comparator)
  Interventions: Device: Standard dialysate (StDi)
- pre-dilution oHDF with citrate dialysate (Experimental)
  Interventions: Device: Citrate dialysate (CiDi)
- HD treated with citrate dialysate (Experimental)
  Interventions: Device: Citrate dialysate (CiDi)
- post-dilution oHDF with citrate dialysate (Experimental)
  Interventions: Device: Citrate dialysate (CiDi)
- pre-dilution oHDF with standard dialysate (Active Comparator)
  Interventions: Device: Standard dialysate (StDi)

INTERVENTIONS:
Device: Citrate dialysate (CiDi) — Use during chronic dialysis 3x/week
  Arms: HD treated with citrate dialysate; post-dilution oHDF with citrate dialysate; pre-dilution oHDF with citrate dialysate
Device: Standard dialysate (StDi) — Use during chronic dialysis 3x/week
  Arms: HD treated with standard dialysate; post-dilution oHDF with standard dialysate; pre-dilution oHDF with standard dialysate

SUMMARY:
Study investigating the safety and efficacy of the citrate dialysis solution compared to standard acetate dialysis solution. Use of citrate dialysis solution is not associated with a clinically relevant development of adverse events. It is hypothesized that citrate dialysate may provide a local anticoagulation effect in the dialyser improving removal of uremic toxins.

DETAILED DESCRIPTION:
It is hypothesized that citrate dialysate may provide a local anticoagulation effect in the dialyser improving removal of uremic toxins. Study investigating the safety and efficacy of the citrate dialysis solution compared to standard acetate dialysis solution. Use of citrate dialysis solution is not associated with a clinically relevant development of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* patients of either sex aged ≥ 18 years
* stable chronic dialysis patients undergoing a 3x/week high-flux dialysis for at least three months
* patients without planned or predictable changes within diet, anticoagulation and medication regimen

Exclusion Criteria:

* pregnancy or lactation or woman in child bearing age without effective contraception
* planned surgeries or hospital stay within the next 9 weeks
* use of catheter as vascular access for dialysis
* severe comorbidities not allowing to follow the study protocol
* concomitant participation in another study
* previous participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2011-10; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of clinically relevant calcium disturbances | patients are followed for 8 weeks
  during or post-dialysis hypocalcaemia with ionized Ca ≤ 0.9 mmol/l
Occurrence of clinically relevant acid-base disturbances | patients are followed for 8 weeks
  during or post-dialysis severe alkalosis with pH ≥ 7.55

SECONDARY OUTCOMES:
Occurrence of clinically relevant acid-base disturbances | patients are followed for 8 weeks
  post-dialysis bicarbonate concentration ≥ 32 mmol/l
Occurrence of clinically relevant acid-base disturbances | patients are followed for 8 weeks
  pre-treatment bicarbonate concentration ≥ 27 mmol/l
Occurrence of clinically relevant intradialytic complications (adverse events) | patients are followed for 8 weeks
  related to citrate dialysate
Occurrence of clinically relevant adverse events | patients are followed for 8 weeks
  related to citrate

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schmitz, Dr., Principal Investigator — Städt. Klinikum Solingen gemeinnützige GmbH Klinik für Nephrologie und Allgemeine Innere Medizin; Olaf Loke, Dr., Principal Investigator — Nephrologische Gemeinschaftspraxis; Klaus Kalb, Dr., Principal Investigator — Märkische Dialysezentren GmbH; Bernhard Fach, Dr., Principal Investigator — PHV Dialysezentrum
Locations (4):
- Germany (4):
  - Märkische Dialysezentren GmbH, Lüdenscheid
  - Nephrologische Gemeinschaftspraxis, Lüdenscheid
  - Städt. Klinikum Solingen gemeinnützige GmbH Klinik für Nephrologie und Allgemeine Innere Medizin, Solingen
  - PHV Dialysezentrum, Wetzlar

REFERENCES:
- [Derived] Natale P, Ju A, Strippoli GF, Craig JC, Saglimbene VM, Unruh ML, Stallone G, Jaure A. Interventions for fatigue in people with kidney failure requiring dialysis. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD013074. doi: 10.1002/14651858.CD013074.pub2. PMID 37651553